CLINICAL TRIAL: NCT05499065
Title: Real-time Margin Assessment in Head and Neck Cancer - Enhancing Specificity by Combining Fresh Frozen Sectioning With Targeted Fluorescence Imaging
Brief Title: Real-time Margin Assessment in Head and Neck Cancer
Acronym: LIGHTNING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Max J.H. Witjes, Prof. dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10968
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: Cetuximab-800CW; Fluorescence guided surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 75mg cetuximab + 15mg cetuximab-800CW (Experimental): To investigate if study drugs can assist in tumor-positive margin detection
  Interventions: Procedure: Fluorescence guided detection of tumor positive margins; Drug: Cetuximab-IRDye800

INTERVENTIONS:
Procedure: Fluorescence guided detection of tumor positive margins — To test if the fluorescence can guide the location for fresh frozen section sampling intra-operatively
Drug: Cetuximab-IRDye800 — Administrate 75mg cetuximab + 15mg cetuximab-800CW for fluorescence visualization

SUMMARY:
To investigate if the combination of fresh frozen sectioning based on cetuximab-800CW can enhance tumor-positive margin detection intra-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Cytology and/or histology-confirmed diagnosis of oral squamous cell carcinoma and scheduled to undergo surgical removal as decided by the multidisciplinary head and neck tumor board of the UMCG;
* Age ≥ 18 years;
* Written informed consent.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Concurrent uncontrolled medical conditions;
* Received an investigational drug within 30 days prior to the dose of cetuximab-800CW;
* History of myocardial infarction, cerebrovascular accident, uncontrolled cardiac heart failure, significant liver disease (ALT >3X upper limits of normal or increased total bilirubin) or unstable angina within 6 months prior to enrollment;
* Inadequately controlled hypertension with or without current antihypertensive medications;
* History of allergy or infusion reactions cetuximab or other monoclonal antibody therapies;
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for women of childbearing potential. Moreover, the need to be willing to ensure that she or her partner uses effective contraception during the trial and for 6 months thereafter. Woman of childbearing potential are premenopausal women with intact reproductive organs and women less than two years after menopause;
* Evidence of QT prolongation on pretreatment ECG (greater than 440 ms in males or greater than 450 ms in females)
* Patients receiving Class 1a (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
* Life expectancy < 12 weeks;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Enhanced intra-operative margin detection | Postoperatively, i.e. 7-10 working days
  To determine the feasibility of fluorescence imaging combined with fresh frozen sectioning of a fluorescence guided biopsy of the excised tissue specimen in an on-site intra-operative setting.
  Outcome parameter: Detection rate of tumor-positive margins based on standard of care histopathological H/E assessment compared to fresh-frozen section analysis combined with fluorescence

CONTACTS AND LOCATIONS:
Overall Officials: Floris J Voskuil, MD, PhD, Principal Investigator — University Medical Center Groningen; Max JH Witjes, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No